CLINICAL TRIAL: NCT02088047
Title: The Effects of ProFoveate on Reducing Self-Stimulating Behaviors in Children Diagnosed With Autism Spectrum Disorders
Brief Title: The Effects of ProFoveate on Reducing Self-Stimulating Behaviors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided to end the study
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202241
Record Dates: First submitted 2014-03-10; First posted 2014-03-14 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Autism Spectrum Disorders; Normal Hearing; Normal Intelligence; Exhibit Self- Stimulating or Ritualistic Behaviors
Keywords: Autism; Self-Stimulating behaviors; Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Profoveate (Experimental): The experimental group will receive the ProFoveate™ intervention along with pre (baseline) and post (end line)intervention assessment. Steel pellets (1.2 mm) will be placed strategically on ears following instructions on how to use the ProFoveate™ pellets. Parents will be provided with a Patient Diary Sheet and will be instructed to perform and document daily checks for placement of the pellets. Parents will be given a one month supply of stainless steel pellets at the initial study visit. Child participants will wear the stainless steel ProFoveate™ pellets for four weeks.
  Interventions: Device: ProFoveate
- NonProFoveate (No Intervention): Participants in the control group will have no intervention. They will receive the initial pre testing (baseline) followed by post testing after 4 weeks.

INTERVENTIONS:
Device: ProFoveate — ProFoveate™ intervention for nystagmus is a management approach comprised of non-magnetic, 1.2 mm spheres that can be made from either stainless steel, gold plated stainless steel or titanium, placed strategically about the face and ears and a set of exercises designed to support improved vision for patients with nystagmus.The spheres (i.e., stimulating press balls or pellets) are supplied in packages of 20 with each sphere supplied on a transparent hypoallergenic adhesive tape approximately 7.6 mm in diameter. Within each package, all spheres are individually contained on a single paper backing measuring approximately 8.5 cm by 1.7 cm. Individual pellets (with adhesive tape) are removed from the backing as needed according to the prescribed treatment regimen.
  Arms: Profoveate

SUMMARY:
This study is designed to pilot an intervention technique to reduce the self-stimulating behaviors seen in individuals with autism spectrum disorders using intervention with ProFoveate pellets. Self-stimulating behaviors like hand flapping, eye blinking, and rocking, can interfere with the individual's ability to interact with their peers. Participants will wear the pellets for four week and measures with taken again. Another group of participants will not get the pellets. Both groups will be tested at the beginning and end of the study. Any variations in self-stimulating behaviors will be documented through parent report, Observational data. The investigators hypothesize that they will see changes in self- stimulating behaviors as a result of the strategic placement of the ProFoveate™ pellets on the ears of one group of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented diagnosis of high functioning autism spectrum disorders (autism, Asperger's syndrome, or Pervasive Development Disorder (PDD) as reported by specialists who use the established criteria (American Psychiatric Association,2000)
* Pass a hearing screening at 25 decibels for the frequencies 1000, 2000 and 4000 hertz
* Score 85 or above on the Test of Nonverbal Intelligence- 4 (TONI-4; Brown, Sherbenou & Johnsen, 2009)
* Exhibit noticeable self- stimulating or ritualistic behaviors (i.e., scratching, hand flapping, eye blinks, etc.) and/or visual characteristics of Autism Spectrum Disorder (ASD) (sensitivity to light, visual fixations, poor eye contact, etc.) as reported by parents and/or observed on videos taken during assessment.

Exclusion Criteria:

* Known history of latex allergy
* Intelligence Score below 85
* Fail the hearing screening

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2014-08-30 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Atcherson, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas at Little Rock Speech and Hearing Clinic, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Profoveate: The experimental group will receive the ProFoveate™ intervention along with pre (baseline) and post (end line)intervention assessment.
Period: Overall Study
Arm/Group | Profoveate | NonProFoveate
Started | 3 | 1
Completed | 2 | 1
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Profoveate | NonProFoveate | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 0 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Self-stimulating Behaviors
Description: Only 4 participants completed enrollment.Only 3 participants completed study. Study was terminated due to low enrollment.
Time Frame: Baseline to 4 Weeks
Population: Students were given a Social Skills Improvement System (SSiS). Only 4 participants completed enrollment. Only 3 participants completed study. Study was terminated due to low enrollment.
Measure: Mean (Standard Deviation); unit: behaviors
Arm/Group | Profoveate | NonProFoveate
Number analyzed (Participants) | 3 | 1
behaviors | 40 (7.24) | 27 (1.6)

ADVERSE EVENTS:
Time Frame: adverse event data was collected for 30 days
Arm/Group | Profoveate | NonProFoveate
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2014-09-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT02088047/Prot_001.pdf